CLINICAL TRIAL: NCT02575430
Title: Retrospective, Uncontrolled, Multicenter, Case History Study to Determine the Natural History of Visual Function in Subjects With Inherited Retinal Disease (IRD) Caused by Inherited Mutation of Retinal Pigment Epithelial 65 Protein (RPE65) or Lecithin:Retinol Acyltransferase (LRAT)
Brief Title: Natural History Study in Inherited Retinal Disease Subjects Caused by Mutations in RPE65 or LRAT
Status: Completed | Type: Observational
Sponsor: QLT Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RET NAT 01
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Leber Congenital Amaurosis (LCA); Retinitis Pigmentosa (RP)
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinitis Pigmentosa

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with IRD: IRD phenotypically diagnosed as Leber congenital amaurosis (LCA) or retinitis pigmentosa (RP) caused by RPE65 or LRAT gene mutations.
  Interventions: Other: No treatment: retrospective chart review

INTERVENTIONS:
Other: No treatment: retrospective chart review

SUMMARY:
To evaluate the natural history of visual function in subjects with IRD phenotypically diagnosed as Leber congenital amaurosis (LCA) or retinitis pigmentosa (RP) caused by RPE65 or LRAT gene mutations.

DETAILED DESCRIPTION:
This is a retrospective, uncontrolled, multicenter, case history study to determine the natural history of visual function in patients with IRD phenotypically diagnosed as LCA or RP caused by autosomal recessive mutation in RPE65 or LRAT.

Up to 60 subjects will be enrolled in this study at approximately 12 study centers in Canada, the US and Europe.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 8 or older with IRD (LCA or RP) caused by inherited autosomal recessive mutation in either RPE65 or LRAT.
* Subjects who have at least 2 documented kinetic visual field assessments of the same isopter(s) in at least one eye performed at least 2 years apart on the same type of equipment when the subject was between the ages of 6 and 65 years.
* If applicable, subjects who provide informed consent for the study (the requirement for informed consent may be applicable to all sites or may be waived by the IRB and/or local regulations). The parent or guardian must sign an approved informed consent form for the study for subjects younger than the age of majority.

Exclusion Criteria:

* Subjects, who in the Investigator's opinion, have any severe acute or chronic medical condition, psychiatric condition, physical examination finding or laboratory abnormality that may interfere with the interpretation of their visual function data.
* Subjects with concomitant bilateral ocular disorders that may affect visual acuity or visual fields (e.g., advanced glaucoma, optic neuritis, anterior ischemic optic neuropathy, advanced cataract, intraocular surgery).

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with IRD phenotypically diagnosed as LCA or RP caused by autosomal recessive mutation in RPE65 or LRAT.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Visual field | Change in visual field over time. Previous assessments performed when subject was between the ages of 6 and 65 years

SECONDARY OUTCOMES:
Visual acuity | Change in visual acuity over time. Previous assessments performed when subject was between the ages of 6 and 65 years

OTHER OUTCOMES:
Optical coherence tomography, if available | Previous assessments performed when subject was between the ages of 6 and 65 years
Electroretinogram, if available | Previous assessments performed when subject was between the ages of 6 and 65 years

CONTACTS AND LOCATIONS:
Overall Officials: David Saperstein, MD, Study Director — QLT Inc.
Locations (9):
- United States (2):
  - Wilmer Eye Institute - Johns Hopkins Hospital, Baltimore, Maryland
  - Casey Eye Institute - Marquam Hill, Portland, Oregon
- Canada (2):
  - The Hospital for Sick Children, Ophthalmology and Vision Sciences, Toronto, Ontario
  - Montreal Children's Hospital, McGill University Health Centre, Montreal, Quebec
- Glostrup Hospital and National Eye Clinic at the Kennedy Center, Glostrup Municipality, Copenhagen, Denmark
- STZ Eyetrial at the Department of Ophthalmology - University of Tübingen, Tübingen, Germany
- Rotterdam Ophthalmic Institute, Rotterdam, Netherlands
- Jules Gonin Eye Hospital - Oculogenetic Unit, Lausanne, Switzerland
- Moorfields Eye Hospital - Research and Treatment Centre, London, United Kingdom